CLINICAL TRIAL: NCT06717100
Title: A Phase 1 Study in Healthy Volunteers to Determine the Potential for Drug-drug Interactions When Co-administering Deupirfenidone (LYT-100) With Nintedanib
Brief Title: Study to Determine Potential for Drug-drug Interactions When Co-administering Deupirfenidone (LYT-100) and Nintedanib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PureTech (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LYT-100-2024-03
Record Dates: First submitted 2024-11-20; First posted 2024-12-04 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Drug Interactions
Keywords: LYT-100; nintedanib; deupirfenidone; drug interaction; interaction; Pulmonary Fibrosis; Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Pulmonary Fibrosis; Idiopathic Pulmonary Fibrosis | interventions — nintedanib; pirfenidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- DDI Cohort (Experimental): All participants will receive the same interventions at the same schedule
  Interventions: Drug: Nintedanib 150 MG [Ofev]

INTERVENTIONS:
Drug: Nintedanib 150 MG [Ofev] — Nintedanib 150 MG will be administered every 12 hours from Days 1 to 20. LYT-100 will be titrated from 275 MG three times a day on Days 8 to 10, to 550 MG three times a day on Days 11 to 13, to 825 MG three times a day on Days 14 to 30.
  Other Names: Deupirfenidone (LYT-100) 275 MG

SUMMARY:
This is a trial of up to 60-day duration for safety, tolerability, and pharmacokinetics in healthy volunteers administered deupirfenidone (LYT-100) alone or in combination with nintedanib .

DETAILED DESCRIPTION:
The purpose of this research is to investigate the effects of deupirfenidone (LYT-100) when co-administered with nintedanib to determine if there are any drug-drug interactions. In particular, the study will investigate the safety, tolerability and pharmacokinetics of LYT-100 co-administered with nintedanib. Eligible participants will be admitted to the Clinical Research Unit for 31 days, will be administered nintedanib and/or LYT-100 for 30 days, and will provide blood samples and have assessments during this time. Participants will return for a safety follow-up visit 30 days after taking the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Provides written Ethics Committee approved informed consent prior to any study procedures.
2. Male or female between 18 and 65 years old (inclusive) at the time of Screening.
3. In good general health at Screening, free from clinically significant unstable and/or acute medical, surgical or psychiatric illness/es and a full physical examination, at the discretion of the Investigator.
4. Clinical laboratory analytes at Screening and Day -1 (including hematology, biochemistry, coagulation, and urinalysis) within normal range as specified by the testing laboratory, unless deemed not clinically significant by the PI.
5. Subjects have a body mass index (BMI) between ≥ 18.0 and ≤ 35.0 kg/m2 and weigh at least 50 kg at Screening.
6. Vital signs (measured in sitting position after 5 minutes' rest) at Screening and at Day -1:

   1. Systolic blood pressure ≥90 and ≤140 mmHg; and
   2. Diastolic blood pressure ≥40 and ≤ 90 mmHg; and
   3. Heart rate ≥40 and ≤100 beats per minute (bpm). Note: If vital signs are out of range, the Investigator may obtain one additional reading, so that up to 2 consecutive assessments are made within 1 hour and with the subject seated quietly during the 5 minutes preceding the assessment.
7. Adequate venous access in the left or right arm to allow collection of multiple blood samples.
8. No relevant dietary restrictions, and willing to consume the entirety of the standard meals provided.
9. Willing to comply with all study procedures and requirements.
10. Willing to abstain from direct whole body sun exposure from 2 days prior to dosing and until EOS/Follow-up Visit.
11. Women of childbearing potential (WOCBP) must be non-pregnant and non-lactating, and must use acceptable, highly effective contraception or be abstinent from heterosexual intercourse if this is their usual sexual practice from Screening until study completion, including the follow-up period and an additional 90 days after the last dose of study drug. Effective forms of contraception are defined in Section 4.4.4 of the protocol. WOCBP must have a negative serum pregnancy test at Screening and negative urine pregnancy test at Day -1 and be willing to have additional pregnancy tests as required throughout the study.
12. Women not of childbearing potential must be post menopausal for ≥12 months (without an alternative medical cause) or be surgically sterile (for which acceptable methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy). Post-menopausal status will be confirmed through testing of follicle stimulating hormone (FSH) levels ≥ 40 IU/L at Screening. Bilateral tubal ligation is acceptable (if completed successfully and done at least one year prior to Screening [verbal confirmation is permitted]), but condom use by male partner is required until study completion including the follow-up period.
13. Male subjects must be surgically sterile (> 90 days since vasectomy with no viable sperm confirmed by laboratory documentation), abstinent if this is their usual sexual practice, or if engaged in sexual relations with a WOCBP, the subject and his partner must be surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy) or using an acceptable, highly effective contraceptive method (See Section 4.4.4 of the protocol) from Screening until study completion, including the follow-up period and an additional 90 days after the last dose of study drug. Male subjects that have undergone a vasectomy must use a condom from Screening until study completion, including the follow-up period and an additional 90 days after the last dose of study drug.
14. Males must not donate sperm and females must not donate ova or oocytes (i.e., human eggs) for at least 90 days after the last dose of study drug.
15. Subjects with same-sex partners (abstinence from penile-vaginal intercourse) or who are abstinent from heterosexual intercourse are not required to use contraception when this is their preferred and usual lifestyle.

Exclusion Criteria:

1. Pregnant or lactating at Screening or Day -1 or planning to become pregnant (self or partner) at any time during the study, including the specified follow-up period.
2. History or presence of malignancy at Screening or Day -1, with the exception of adequately treated localised skin cancer (basal cell or squamous cell carcinoma) or carcinoma in-situ of the cervix.
3. History of migraine, whether treated or untreated, within 3 years prior to Screening
4. Clinically significant infection within 28 days of the start of dosing, or infections requiring parenteral antibiotics within the 6 months prior to Screening.
5. Clinically significant surgical procedure within 3 months of Screening, at the discretion of the Investigator, or any planned significant surgical procedure prior to the EOS/Follow-up visit.
6. Family history (biological relatives [i.e., parents, siblings]) of long or short QT syndrome, or Torsades de Pointes.
7. Currently suffering from clinically significant systemic allergic disease at Screening or Day -1 or has a history of significant drug allergies including a history of anaphylactic reaction; allergic reaction due to any drug which led to significant morbidity; prior allergic reaction to pirfenidone.
8. Chronic administration (defined as more than 14 consecutive days) of immunosuppressants or other immune-modifying drugs within 3 months prior to study drug administration; corticosteroids are permitted at the discretion of the Investigator). Topical agents are not exclusionary.
9. History or presence at Screening or Day -1 of a condition associated with significant immunosuppression.
10. Positive result of a RT-qPCR diagnostic test for SARS-CoV-2 at Screening or Day -1.
11. Positive test for hepatitis C antibody (HCV), hepatitis B surface antigen (HBsAg), or human immunodeficiency virus (HIV) antibody at Screening. Subjects who are positive for HCVAb will be tested for hepatitis C ribonucleic acid (HCV RNA) by polymerase chain reaction (PCR) and, if HCV RNA PCR is positive, will be excluded.
12. Symptoms of dysphagia at Screening or Day -1 or known difficulty in swallowing capsules.
13. History or presence of gastrointestinal (including a previous episode of pancreatitis), hepatic or renal disease, or any other conditions known to interfere with absorption, distribution, metabolism, or excretion of drugs.
14. Any condition at Screening or Day -1 (e.g., chronic diarrhoea, inflammatory bowel disease or prior surgery of the gastrointestinal tract) that would interfere with drug absorption or any disease or condition that is likely to affect drug metabolism or excretion, at the discretion of the Investigator.
15. History or presence at Screening or Day -1 of cardiac arrhythmia or congenital long QT syndrome.
16. QT interval corrected using Fridericia's formula (QTcF) > 450 msec (male) or 470 msec (female) demonstrated by two ECGs 30 to 60 minutes apart at Screening or Day -1 visits. The average of the 2 QTcF intervals should be used to determine the subject's eligibility.
17. Use of smoked tobacco or nicotine containing products in the previous 3 months prior to dosing or use of other tobacco or nicotine containing products in the previous 2 weeks prior to dosing, or a positive urine cotinine test at Screening or Day -1.
18. Lack of willingness to abstain from the consumption of tobacco or nicotine-containing products throughout the duration of the study and until the EOS/Follow-up visit.
19. Lack of willingness to abstain from the use of alcohol throughout the study (Treatment through EOS/Follow-up visit).
20. Positive toxicology screening panel (urine test, including qualitative identification of barbiturates, tetrahydrocannabinol [THC], amphetamines, benzodiazepines, opiates and cocaine) or alcohol breath test at Screening or Day -1, at any time during the Study. One repeat urine toxicology screen may be conducted, within 48 h of the first, if the first is considered by the Investigator to be invalid.
21. History of substance abuse or dependency or history of recreational intravenous (IV) drug use, over the last 2 years.
22. Use of any prescription drugs, over the counter (OTC) medication, nonsteroidal anti-inflammatory agents (NSAIDs), herbal remedies, supplements or vitamins within the 14 days prior to dosing or throughout the duration of the study, without prior approval of the Investigator and written approval of the Medical Monitor.
23. Paracetamol/acetaminophen may be utilised, provided that the dose of paracetamol does not exceed 2 g in any 24 h period.
24. Use of any of the any drugs listed in Section 4.4.1 within 28 days or 5 half-lives of that drug, whichever is longer, prior to study drug administration.
25. Vaccination with a live vaccine within the 4 weeks prior to Screening or that is planned prior to the EOS visit, and any non-live vaccination within the 2 weeks prior to Screening or that is planned within 2 weeks of dosing (including those for COVID-19)
26. Exposure to any significantly immune suppressing drug within the 3 months prior to Screening or 5 half lives, whichever is longer.
27. Use of any investigational drug or device within 3 months prior to Screening.
28. Consumption of soy, grapefruit, grapefruit juice, Seville oranges, Seville orange juice, or any foods containing these ingredients, within 7 days prior to dosing until 24 hours after the final dose of study drug or unwilling to abstain from these throughout the duration of the study, until the EOS visit.
29. Clinically significant blood loss, blood or blood product donation >250 mL within 28 days of Screening.
30. Subject is unwilling to refrain from strenuous exercise which significantly exceeds the subject's usual level of physical activity from 48 h prior to admission to the clinical trial unit and until completion of the final onsite follow-up visit, where strenuous exercise is defined as a significant increase in the Subject's usual level of physical activity or lifting weights or running uphill.
31. Any other reason that, in the opinion of the Investigator, might interfere with the evaluation required by the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-12-17 (Actual); Primary Completion 2025-02-17 (Actual); Study Completion 2025-03-17 (Actual)

PRIMARY OUTCOMES:
AUC of LYT-100 and nintedanib | 0-tlast: Day 1 to 20 for nintedanib; Day 8 to 30 for LYT-100
  The area under the curve will be calculated from the first observed to last measurable plasma concentration. For nintedanib, dosing begins on Day 1 and ends on Day 20. For LYT-100, dosing begins on Day 8 and ends on Day 30.
AUC of LYT-100 and nintedanib | 0-12 hour
AUC of LYT-100 | 0-6 hour
Tmax of LYT-100 and nintedanib | 0-12 hour
Cmax of LYT-100 and nintedanib | 0-12 hour

SECONDARY OUTCOMES:
Adverse Events | Screening through Follow-up Visit on Day 60
  Adverse events defined as an untoward medical occurrence that occurs in conjunction with the use of a medicinal product in humans, whether or not considered to have a causal relationship to this treatment will be recorded and followed. Description, duration, causality, severity, seriousness, actions taken, and outcomes for all adverse events will be reported and analyzed.
Number of subjects with abnormal vital signs (blood pressure) | Screening through Follow-up Visit on Day 60
  Systolic and Diastolic blood pressure measured in millimeters of mercury (mmHg)
Number of subjects with abnormal vital signs (heart rate) | Screening through Follow-up Visit on Day 60
  Heart rate measured in beats per minute (bpm)
Number of subjects with abnormal vital signs (respiration rate) | Screening through Follow-up Visit on Day 60
  Respiration rate measured in breaths per minute (bpm)
Number of subjects with abnormal vital signs (body temperature) | Screening through Follow-up Visit on Day 60
  Tympanic body temperature measured in degrees Celsius
Number of subjects with abnormal vital signs (oxygen saturation) | Screening through Follow-up Visit on Day 60
  Oxygen saturation measured in percentage
Number of subjects with abnormal electrocardiograms | Screening through Follow-up Visit on Day 60
Number of subjects with abnormal physical examinations | Screening through Follow-up Visit on Day 60
Number of subjects with abnormal laboratory values (hematology) | Screening through Follow-up Visit on Day 60
  Hematology parameters to be tested are hemoglobin, hematocrit, erythrocytes, platelets, and leukocytes.
Number of subjects with abnormal laboratory values (serum chemistry) | Screening through Follow-up Visit on Day 60
  Serum chemistry parameters to be tested are C-reactive protein, urea, creatinine, total and direct bilirubin, urate, albumin, globulin, alkaline phosphatase, creatine phosphokinase, troponin 1, aspartate aminotransferase, alanine aminotransferase, gamma-glutamyl transpeptidase, glucose, sodium, potassium, calcium, chloride, phosphate, bicarbonate
Number of subjects with abnormal laboratory values (coagulation) | Screening through Follow-up Visit on Day 60
  Coagulation parameters to be tested are international normalized ratio, prothrombin time, activated partial thromboplastin time
Number of subjects with abnormal laboratory values (urinalysis) | Screening through Follow-up Visit on Day 60
  Urinalysis parameters to be tested are micro protein, nitrite, pH, trial specific gravity, ketone bodies, urobilinogen, blood, urine leukocyte esterase, appearance uri acm, micro glucose, bilirubin

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network Pty Ltd (Commercial Rd and St Kilda Rd) - VIC, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No